CLINICAL TRIAL: NCT00199641
Title: Evaluation of Two Enteral Nutrition Strategies in Mechanically Ventilated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DGS 2002/0361
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2008-12-04 (Estimated); Status verified 2008-12

CONDITIONS: -Mechanically Ventilated Patients
MeSH Terms: interventions — Enteral Nutrition

INTERVENTIONS:
Device: enteral nutrition

SUMMARY:
The aim of this study is to compare two strategies of early enteral nutrition in terms of efficacy and complications in mechanically ventilated patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 18 ans)
* Mechanical ventilation for > 72 hours
* Planned enteral nutrition
* Informed consent

Exclusion Criteria:

* Body Mass Index < 20 kg/m2
* Enteral nutrition non indicated (ileus, splanchnic ischemia..)
* Shock (use of catecholamines, arterial blood pressure < 90 mmHg, peripheral hypoperfusion, elevation of lactates > x 1,5 normal value)
* Contraindications for gastric tube
* Pregnancy
* Previous enrollment in the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2002-07

PRIMARY OUTCOMES:
Incidence of nutrition failure (diarrhea, ileus, vomiting, aspiration pneumonia, elevated residual gastric volume)

SECONDARY OUTCOMES:
-Measured nutrition amount when compared to theorical nutrition during ICU stay
-Measured nutrition amount when compared to theorical nutrition during the first three days
-Influence of prokinetic drugs on nutrition quality

CONTACTS AND LOCATIONS:
Overall Officials: Bruno François, MD, Principal Investigator — University Hospital, Limoges
Locations (2):
- France (2):
  - Service de Réanimation, Angoulême
  - Service de réanimation Polyvalente, Limoges